CLINICAL TRIAL: NCT05893589
Title: The Impact of the Social Cognitive Theory Based Educational Program on Women-headed Households' Social Health : A Field Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gonabad University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Atefeh Dehnoalian, Social Development and Health Promotion Research Center, Gonabad University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IR.GMU.REC.1398.172
Record Dates: First submitted 2023-05-07; First posted 2023-06-08 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-05

CONDITIONS: Social Behavior; Health Behavior
MeSH Terms: conditions — Social Behavior; Health Behavior

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- test (Experimental)
  Interventions: Other: test group
- control group (No Intervention)

INTERVENTIONS:
Other: test group — Women in the intervention group participated in face-to-face and virtual meetings based on social cognitive theory structures for 4 weeks
  Arms: test

SUMMARY:
The goal of this field trial was to compare in emale-headed households. The main question it aims to answer are:

determine the effect of education based on social cognitive theory on the social health of female-headed households in female-headed households in Gonabad.

Women in the intervention group participated in face-to-face and virtual meetings based on social cognitive theory structures for 4 weeks. The control group did not receive any training related to the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent to participate in the study, being the head of the household, age range from 20 to 64 years, ability to speak and listen, reading and writing literacy, access to a mobile phone with Android operating system to receive educational messages (access to the Internet and virtual networks) or Having access to a person who will help him in using virtual networks, not suffering from acute diseases and hospitalization during the intervention.

Exclusion Criteria:

* Dissatisfaction to continue cooperation, not completing the questionnaire completely

Ages: 20 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2021-05-10 (Actual); Primary Completion 2021-05-10 (Actual); Study Completion 2022-05-20 (Actual)

PRIMARY OUTCOMES:
social health | before
  Social health is measured by the Keyes Social Health Questionnaire. This questionnaire
social health | After 4 weeks
  Social health is measured by the Keyes Social Health Questionnaire. This questionnaire includes 20 questions and examines 5 subscales of social prosperity, social solidarity, social cohesion, social acceptance and social participation.relationships with others

CONTACTS AND LOCATIONS:
Locations (1):
- A;ian, Neyshabur, Khorasan Razavi, Iran

IPD SHARING:
Plan to Share IPD: No